CLINICAL TRIAL: NCT03006562
Title: A Randomized Controlled Trial for PREvention of VENous ThromboEmbolism Following Radical Prostatectomy (PREVENTER Trial)
Brief Title: PREvention of VENous ThromboEmbolism Following Radical Prostatectomy
Acronym: PREVENTER
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early stopping point based on 2nd interim analysis (planned per protocol)
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00123618
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer; Venous Thromboembolism; Lymphocele After Surgical Procedure; Deep Venous Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Prostatic Neoplasms; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Prospective, single-institution, multi-surgeon, stratified randomized controlled trial. Randomization will be stratified into four groups by procedure approach (open or robotic) and whether patients elect to undergo a screening 30-day lower extremity Duplex (ultrasound or no ultrasound). Patients will then be randomized, within each of the strata, to the two arms (subcutaneous heparin versus no subcutaneous heparin).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subcutaneous Heparin (Experimental): Patients randomized to the pharmacologic VTE prophylaxis arm will receive a dose of subcutaneous heparin 5,000 units prior to incision, and subcutaneous heparin 5,000 units every 8 hours after surgery until discharge.
  Interventions: Drug: Subcutaneous Heparin
- Control (No Intervention): Patients randomized to the control arm will receive routine care with intermittent pneumatic compression devices.

INTERVENTIONS:
Drug: Subcutaneous Heparin — 5,000 units of subcutaneous heparin before surgery and then every 8 hours after surgery until discharge from the hospital.
  Arms: Subcutaneous Heparin

SUMMARY:
The PREVENTER Trial aims to compare the use of perioperative pharmacologic prophylaxis (subcutaneous heparin) with intermittent pneumatic compression devices (IPCs) to the use of IPCs alone for the prevention of venous thromboembolism (VTE) after radical prostatectomy (RP).

DETAILED DESCRIPTION:
The PREVENTER Trial aims to compare the use of perioperative pharmacologic prophylaxis (subcutaneous heparin) with intermittent pneumatic compression devices (IPCs) to the use of IPCs alone for the prevention of venous thromboembolism (VTE) after radical prostatectomy (RP). Currently, there is no standard practice for VTE prophylaxis after RP with the American Urological Association recommending "pharmacological or pneumatic mechanical prophylaxis" for high risk patients. Prior studies showed 30% of patients in the United States received no perioperative prophylaxis and less than 20% received pharmacologic agents, compared to 98% of patients receiving pharmacologic prophylaxis in the United Kingdom. Some urologists prescribe patients low molecular weight heparin (LMWH) after discharge for up to 30 days after surgery. Additionally, there are no established risks of pharmacologic prophylaxis for RP patients, but some urologists express concern about the potential impact of prophylaxis on the rate of postoperative lymphoceles or hematomas. At Johns Hopkins, patients do not routinely receive pharmacologic VTE prophylaxis in the perioperative setting for RP. Given the lack of standard practice and implications for patient safety, the investigators propose a prospective, stratified randomized controlled trial to evaluate the impact of perioperative pharmacologic prophylaxis on VTE following RP hypothesizing that it will prevent VTE events without significantly impacting the rate of postoperative bleeding or lymphoceles. The potential impact of surveillance bias with differential imaging between arms, effect of lymphadenectomy (yes/no and number of noted removed) or surgical approach (robotic and open), and differences by patients risk (comorbidity and VTE risk based on components of the Caprini score) or demographics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men 18-100 years of age with histologically confirmed prostate cancer of any stage undergoing RP
* Patients who would have otherwise been eligible to receive routine post-RP care

Exclusion Criteria:

* Active treatment for VTE
* Patients judged by patients' urologist, primary care doctor, or in the preoperative evaluation center (PEC) to be unsafe to forgo pharmacologic prophylaxis or systemic anticoagulation postoperatively (whether or not patients are on systematic anticoagulation for indications other than VTE)
* Known adverse reactions to heparin (heparin-induced thrombocytopenia or any allergy)
* Epidural analgesia
* Spinal anesthesia
* Participation in a different trial that increases a patient's risk of VTE

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad E Allaf, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang MM, Su ZT, Becker REN, Pavlovich CP, Partin AW, Allaf ME, Patel HD. Complications after open and robot-assisted radical prostatectomy and association with postoperative opioid use: an analysis of data from the PREVENTER trial. BJU Int. 2021 Feb;127(2):190-197. doi: 10.1111/bju.15172. Epub 2020 Aug 17. PMID 32654363
- [Result] Patel HD, Faisal FA, Trock BJ, Joice GA, Schwen ZR, Pierorazio PM, Johnson MH, Bivalacqua TJ, Han M, Gorin MA, Carter HB, Partin AW, Pavlovich CP, Allaf ME. Effect of Pharmacologic Prophylaxis on Venous Thromboembolism After Radical Prostatectomy: The PREVENTER Randomized Clinical Trial. Eur Urol. 2020 Sep;78(3):360-368. doi: 10.1016/j.eururo.2020.05.001. Epub 2020 May 19. PMID 32444264
- [Derived] Patel HD, Faisal FA, Patel ND, Pavlovich CP, Allaf ME, Han M, Herati AS. Effect of a prospective opioid reduction intervention on opioid prescribing and use after radical prostatectomy: results of the Opioid Reduction Intervention for Open, Laparoscopic, and Endoscopic Surgery (ORIOLES) Initiative. BJU Int. 2020 Mar;125(3):426-432. doi: 10.1111/bju.14932. Epub 2019 Nov 15. PMID 31643128
- [Derived] Patel HD, Srivastava A, Patel ND, Faisal FA, Ludwig W, Joice GA, Schwen ZR, Allaf ME, Han M, Herati AS. A Prospective Cohort Study of Postdischarge Opioid Practices After Radical Prostatectomy: The ORIOLES Initiative. Eur Urol. 2019 Feb;75(2):215-218. doi: 10.1016/j.eururo.2018.10.013. Epub 2018 Oct 21. PMID 30352714

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subcutaneous Heparin | Control
Started | 251 | 250
Voluntary Ultrasound at 30 Days | 141 | 137
Completed | 251 | 249
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subcutaneous Heparin | Control | Total
Number analyzed (Participants) | 251 | 250 | 501
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [57 to 67] | 61 [56 to 67] | 62 [57 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 251 | 250 | 501
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 200 | 204 | 404
  African American | 34 | 39 | 73
  Hispanic | 8 | 2 | 10
  Asian | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Venous Thromboembolism
Description: Venous thromboembolism (VTE) is a disease that includes both deep vein thrombosis (DVT) and pulmonary embolism (PE). The primary outcome is diagnosis of DVT or PE within 30 days after surgery due to imaging (any method, most commonly lower extremity ultrasound or computed tomography scan with pulmonary embolus protocol) prompted by symptoms of a DVT (lower extremity swelling, pain, fever of unknown origin) or PE (chest pain, shortness of breath, hypoxemia, tachycardia or fever of unknown origin, productive cough with bloody sputum).
Time Frame: 30 days
Population: One participant in the control arm was lost to follow-up precluding outcome assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Heparin | Control
Number analyzed (Participants) | 251 | 249
Participants | 2 | 5

2. Primary Outcome: Number of Participants With Symptomatic Postoperative Fluid Collection
Description: This outcome is defined as a surgical or pelvic fluid collection diagnosed as a hematoma (blood collection, with or without infection) or lymphocele (collection of lymph fluid in the pelvis) due to symptoms (fever, abdominal pain, nausea or vomiting, anemia, high surgical drain output) within 30 days after surgery.
Time Frame: 30 days
Population: One participant in the control arm was lost to follow-up precluding outcome assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Heparin | Control
Number analyzed (Participants) | 251 | 249
Participants | 10 | 9

3. Primary Outcome: Number of Participants With Major Postoperative Bleeding
Description: This additional primary outcome includes the development and diagnosis of any major clinically recognized bleeding event within 30 days after surgery requiring >1 unit of packed red blood cell transfusion, intervention to stop bleeding, or return to the operating room.
Time Frame: 30 days
Population: One participant in the control arm was lost to follow-up precluding outcome assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Heparin | Control
Number analyzed (Participants) | 251 | 249
Participants | 4 | 2

4. Secondary Outcome: Number of Participants With Occurrence of Any Venous Thromboembolism
Description: DVT or PE diagnosed for any reason within 30 days after surgery. This includes any diagnosed DVT or PE as described in the primary outcome plus any additional DVTs or PEs diagnosed at 30 day screening lower extremity ultrasound for patients opting to undergo screening bilateral lower extremity Duplex ultrasound at 30 days who do not have symptoms.
Time Frame: 30 days
Population: Only the subset receiving ultrasound are analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Heparin | Control
Number analyzed (Participants) | 141 | 137
Participants | 4 | 4

5. Secondary Outcome: Estimated Blood Loss During Surgery
Description: The total recorded intraoperative estimated blood loss in milliliters reported at the end of the surgery.
Time Frame: During surgery (usually between 2-3 hours of operative time)
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | Subcutaneous Heparin | Control
Number analyzed (Participants) | 251 | 250
milliliters | 150 [100 to 300] | 200 [100 to 300]

6. Secondary Outcome: Surgical Drain Output After Surgery
Description: The total output in milliliters from any surgical drain left in place (not all patients will necessarily have a surgical drain) after surgery and until discharge from the hospital (usually 1 to 2 days). Drain output, if one is left in place after discharge, will not count toward this secondary outcome.
Time Frame: Over length of stay in hospital (usually 1 to 2 days)
Measure: Median (Inter-Quartile Range); unit: milliliters
Arm/Group | Subcutaneous Heparin | Control
Number analyzed (Participants) | 251 | 250
milliliters | 95 [60 to 180] | 100 [54 to 150]

7. Secondary Outcome: Surveillance Bias by Differential Use of Imaging as Assessed by Number of Participants Receiving Postoperative Diagnostic Imaging for Venous Thromboembolism Relative to Symptoms
Description: Patients in each arm receiving postoperative diagnostic imaging for venous thromboembolism relative to symptoms (e.g. lower extremity Duplex ultrasound, spiral CT angiography, V/Q scan).
Time Frame: 30 days
Population: One participant in the control arm was lost to follow-up precluding outcome assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Heparin | Control
Number analyzed (Participants) | 251 | 249
Participants | 25 | 31

ADVERSE EVENTS:
Time Frame: 30 days
Description: Clavien-Dindo Complications
Arm/Group | Subcutaneous Heparin | Control
All-Cause Mortality (participants affected / at risk) | 0/251 | 0/250
Serious Adverse Events (participants affected / at risk) | 9/251 | 9/250
Other Adverse Events (participants affected / at risk) | 34/251 | 30/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Heparin (N=251) | Control (N=250)
Clavien III or Greater Complication (Surgical and medical procedures) | 9 (9) | 9 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subcutaneous Heparin (N=251) | Control (N=250)
Clavien I or II Complication (Surgical and medical procedures) | 34 (34) | 30 (30)

LIMITATIONS AND CAVEATS:
The study met a futility end point at the 2nd interim analysis (pre-planned in the study protocol) leading to an appropriate decision for early closure and termination rather than continuing to planned enrollment of N=666.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT03006562/Prot_SAP_000.pdf